CLINICAL TRIAL: NCT04909996
Title: Post-market, Confirmatory, Interventional, Randomized and Controlled Clinical Study to Assess the Efficacy and Safety of Sentinox in COVID-19 Patients.
Brief Title: Study on the Performance and Safety of Sentinox in COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: APR Applied Pharma Research s.a. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STX-2021
Record Dates: First submitted 2021-05-28; First posted 2021-06-02 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: COVID-19 (SARS-CoV-2 Infection)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Sentinox treatment performed 3 times/day for 5 days (as add-on to the standard therapy) (Experimental)
  Interventions: Device: Sentinox--Group A
- Group B: Sentinox treatment performed 5 times/day for 5 days (as add-on to the standard therapy) (Experimental)
  Interventions: Device: Sentinox--Group B
- Group C: no Sentinox treatment; only the standard therapy will be performed (No Intervention)

INTERVENTIONS:
Device: Sentinox--Group A — GROUP A: Sentinox treatment performed 3 times/day for 5 days (as addon to the standard therapy) at 8am, 2pm and 8pm;
  The application of IP on should be performed in accordance to the following indication:
  The treatment is administered in a dose of 0.5 ml into each nostril (5 sprays) per the number of times per day according the trial group assigned according the randomization procedure (i.e., GROUP A: 3 times/day; GROUP B: 5 times/day; GROUP C: no IP treatment).
  Arms: Group A: Sentinox treatment performed 3 times/day for 5 days (as add-on to the standard therapy)
Device: Sentinox--Group B — GROUP B: Sentinox treatment performed 5 times/day for 5 days (as addon to the standard therapy) at 8am, 11am, 2pm, 5pm and 8pm;
  The application of IP on should be performed in accordance to the following indication:
  The treatment is administered in a dose of 0.5 ml into each nostril (5 sprays) per the number of times per day according the trial group assigned according the randomization procedure (i.e., GROUP A: 3 times/day; GROUP B: 5 times/day; GROUP C: no IP treatment).
  Arms: Group B: Sentinox treatment performed 5 times/day for 5 days (as add-on to the standard therapy)

SUMMARY:
This is a single-center, randomized, controlled, open-label, pilot study to assess the safety and the performance of Sentinox medical device in the treatment of mild COVID-19 patients.

The study will consist of 9 visits. At the screening visit, according to the investigational site procedures, patients with a positive COVID-19 nasopharyngeal swab (quantitative swab test with RT-PCR Ct value ≤ 30 for at least 2 genes out of 4) performed at the investigational site on the same day will be summoned. Patients will be enrolled after having signed the informed consent form prior to any other study procedure and after inclusion/exclusion criteria check. According to the investigator's judgment, the patient's clinical outcomes, and the investigational site guidelines, the enrolled patients should be hospitalized or redirected to other structures (e.g. "COVID-19 hotel", patient's home).

At Visit 0 (day 0), the patient will be randomized with a 1:1:1 ratio in one of 3 trial groups:

1. Group A: Sentinox treatment performed 3 times/day for 5 days (as add-on to the standard therapy);
2. Group B: Sentinox treatment performed 5 times/day for 5 days (as add-on to the standard therapy);
3. Group C: no Sentinox treatment; only the standard therapy will be performed.

The allocation of the patient in one of the three study arms will be performed sequentially by the principal investigator or delegates in the order in which the subjects are enrolled and will be reported in a randomization list, including the identification code of the patient and the treatment arm (A, B or C) assigned.

At Visit 1 (day 1) and Visit 2 (day 2), three nasopharyngeal swabs will be performed. At subsequent planned visits only one nasopharyngeal swab will be performed in the morning. From Visit 1 (day 1) to Visit 5 (day 5), patients will record daily adverse events (AE), concomitant medication, and presence of clinical features COVID-19 related in a diary.

After the end of the treatment visit (Visit 5), three follow-up visits will be performed on day 6, day 10, and day 21 respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patient Informed consent form (ICF) signed;
* M & F Aged ≥ 18 years and ≤ 64 years at the time of the signature of ICF;
* Subjects who are willing to comply with the requirements of the study protocol, attend scheduled visits and calls for the duration of the study by telephone contact;
* Mild Symptomatic Individuals with COVID-19 confirmed by polymerase chain reaction (PCR) based on WHO guideline (version of 27 May 2020). In the study COVID-19 patient with RT-PCR Ct value ≤ 30 for at least 2 genes out of 4, at the first swab will be enrolled. The enrollment of COVID-19 vaccinated patients will be allowed if they will present a "clinical vaccination failure", defined according to the indications reported in the "Global Manual on Surveillance of AE Following Immunization" (WHO guidelines).
* Onset of symptoms from not more than 2/3 days

Exclusion Criteria:

* Other clinically significant and uncontrolled pathologies that may interfere with study results (e.g. rheumatic diseases);
* Presence of any relevant organic, systemic or metabolic disease (particularly significant history of cardiac, renal, neurological, psychiatric, oncology, endocrinology, metabolic or hepatic disease), or abnormal laboratory values that will be deemed clinically significant based on predefined values;
* Immune system illnesses;
* Known drug and/or alcohol abuse;
* Individuals who are cognitively impaired and/or who are unable to give informed consent;
* Ongoing or prior participation in any other clinical trial of an experimental treatment for COVID-19;
* Ongoing or prior participation in any other clinical trial of an experimental treatment within 30 days from enrollment day;
* Intubated or prior intubation (during present hospitalization) or anticipated intubation within the subsequent 2 hours;
* Using high-flow nasal cannula (HFNC) or non-invasive ventilation (NIV);
* Concurrent or planned treatment with other agents with actual or possible direct antiviral activity;
* Prior hospitalization for COVID-19;
* Positive pregnancy test or breastfeeding woman;*
* Known hypersensitivity to the study treatment, its metabolites, or formulation excipient;
* History of severe drug and / or food allergies and / or known allergies to the trial product or its components;
* Any condition that, in the opinion of the Investigator, would complicate or compromise the study or well-being of the patient.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of Sentinox versus Standard Treatment in term of reduction in viral load (copies/mL) in nasal fluids in mild COVID-19 patients | Day 1,2,3,4 and 5

SECONDARY OUTCOMES:
Efficacy of Sentinox versus Standard Treatment in term of reduction in viral load in nasal fluids in mild COVID-19 patients stratifying the results according to the initial viral load | Day 1,2,3,4,5,6,10 and 21
Time profile of Sentinox to affect the profile of viral load analysing the subjects' negativization (expressed as number of negativized patients) | Day 1,2,3,4,5,6,10 and 21
Time profile of Sentinox to affect the profile of viral load analysing the infectiousness of the patients (expressed as number of infective patients) | Day 1,2,3,4,5,6,10 and 21
To compare the two treatments schedule of Sentinox: 3 irrigations die versus 5 irrigation die in term of reduction in viral load (copies/mL) in nasal fluids | Day 1,2,3,4 and 5
Time profile of Sentinox to affect the profile of viral load (copies/mL) during the duration of the study (treatment period and follow-up period) | Day 1,2,3,4,5,6,10 and 21
Time profile of Sentinox to affect the duration of clinical features of disease using an ad hoc questionnaire during all study duration | Day 1,2,3,4,5,6,10 and 21
Tolerability of the Sentinox a Visual Analogue Scale (VAS) will be used (score 0=not tolerable; score 10=totally tolerable) | Day 6
The patient satisfaction will be evaluated with a 5-points Likert Scale (score 1=not satisfied; score 5=fully satisfied) | Day 6
Safety will be monitored through Adverse Events including assessment of relationship to the IP | Day 1,2,3,4,5,6,10 and 21
Safety will be monitored through clinical examination: difficulty breathing | Day 1,2,3,4,5,6,10 and 21
Safety will be monitored through clinical examination: body temperature | Day 1,2,3,4,5,6,10 and 21
Safety will be monitored through clinical examination: headache | Day 1,2,3,4,5,6,10 and 21
Safety will be monitored through clinical examination: oxygen saturation | Day 1,2,3,4,5,6,10 and 21

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Policlinico San Martino IRCCS, Genova, Italy

REFERENCES:
- [Derived] Panatto D, Orsi A, Bruzzone B, Ricucci V, Fedele G, Reiner G, Giarratana N, Domnich A, Icardi G, Stx Study Group. Efficacy of the Sentinox Spray in Reducing Viral Load in Mild COVID-19 and Its Virucidal Activity against Other Respiratory Viruses: Results of a Randomized Controlled Trial and an In Vitro Study. Viruses. 2022 May 12;14(5):1033. doi: 10.3390/v14051033. PMID 35632774